CLINICAL TRIAL: NCT03023761
Title: Management of Post Endodontic Re-treatment Pain With Low-Level Laser Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University (Other)
Responsible Party: Principal Investigator, saranaz azari-marhabi, assistant professor, Shahid Beheshti University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 123
Record Dates: First submitted 2017-01-11; First posted 2017-01-18 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Pain
Keywords: Endodontic retreatments; Low level laser; Pain
MeSH Terms: conditions — Pain | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- low level laser (Active Comparator): A single visit Endodontic retreatment was done. After biomechanical preparation, Low Level Laser was irradiated to the buccal and lingual mucosa overlying the apices of the target tooth in the experimental group
  Interventions: Device: low level laser
- laser sham (Placebo Comparator): In the control group patients received placebo laser to eliminate the probable psychological effects of laser.
  Interventions: Device: laser sham

INTERVENTIONS:
Device: low level laser — low level laser irradiation
  Arms: low level laser
Device: laser sham — laser without irradiation
  Arms: laser sham

SUMMARY:
In this clinical trial investigators aimed to evaluate Post endodontic re-treatment pain after irradiation of low level laser therapy

DETAILED DESCRIPTION:
In this clinical trial, 61 patients requiring endodontic retreatments in the posterior teeth were selected. A single visit Endodontic retreatment was done. After biomechanical preparation, Low Level Laser was irradiated to the buccal and lingual mucosa overlying the apices of the target tooth in the experimental group. In the control group patients received placebo laser to eliminate the probable psychological effects of laser. Laser irradiation was done with a single dose of 808 nm wavelength (Whitening Lase II- Laser DMC, Samsung, Korea) with 100 mw power, and dose of 70 J/cm2 for 80 seconds. Pain severity was recorded before the treatment, immediately after the treatment and 4, 8, 12, 24 and 48 hours after the treatment by visual analogue scale (VAS). The pain scores were statistically analyzed by chi-square test between two groups. The effects of different variables on the post-operative pain experience were also studied by means of Logistic regression.

ELIGIBILITY:
Inclusion Criteria:

- patients requiring endodontic retreatments in the posterior teeth

Exclusion Criteria:

* systemic diseases psychologic disorders

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 61 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-03 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
reduction of pain after low level laser irradiation | baseline and 4, 8, 12, 24 and 48 hours after the treatment

CONTACTS AND LOCATIONS:
Overall Officials: mohammad asnaashari, Study Chair — Shahid Beheshti University of Medical Sciences
Locations (1):
- Shahid Beheshti University, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Undecided